CLINICAL TRIAL: NCT00539929
Title: Proof of Principle, Randomized, Parallel-Group, Double-Blind, Vehicle-Controlled, Paired-Comparison Study Evaluating the Efficacy and Safety of E6201 Versus Vehicle for the Treatment of Plaque-Type Psoriasis
Brief Title: Paired-Comparison Study Evaluating the Efficacy and Safety of E6201 Versus Vehicle for the Treatment of Plaque-Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E6201-A001-201
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- E6201 0.005% BID (Experimental): Participants applied E6201 0.005% cream to a pre-identified marker lesion twice a day (BID) for 8 weeks. Participants applied matching placebo cream to another pre-identified marker lesion at the same treatment regimen.
  Interventions: Drug: E6201 0.005%; Drug: Placebo
- E6201 0.01% BID (Experimental): Participants applied E6201 0.01% cream to a pre-identified marker lesion BID for 8 weeks. Participants applied matching placebo cream to another pre-identified marker lesion at the same treatment regimen.
  Interventions: Drug: E6201 0.01%; Drug: Placebo
- E6201 0.03% BID (Experimental): Participants applied E6201 0.03% cream to a pre-identified marker lesion BID for 8 weeks. Participants applied matching placebo cream to another pre-identified marker lesion at the same treatment regimen.
  Interventions: Drug: E6201 0.03%; Drug: Placebo
- E6201 0.03% QD (Experimental): Participants applied E6201 0.03% cream to a pre-identified marker lesion once a day (QD) for 8 weeks. Participants applied matching placebo cream to another pre-identified marker lesion at the same treatment regimen.
  Interventions: Drug: E6201 0.03%; Drug: Placebo

INTERVENTIONS:
Drug: E6201 0.005%
  Arms: E6201 0.005% BID
Drug: E6201 0.01%
  Arms: E6201 0.01% BID
Drug: E6201 0.03%
  Arms: E6201 0.03% BID; E6201 0.03% QD
Drug: Placebo

SUMMARY:
This is a double-blind, multicenter study to assess the efficacy and safety of E6201 topical administration to pre-identified marker lesions in adult subjects with chronic plaque type psoriasis. Treatment duration is 8 weeks, followed by a 4-week period without treatment. Pharmacokinetic samples will be obtained pre-and post treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Males and females 18 years or older with a clinical diagnosis of mild-to-moderate plaque-type psoriasis for ≥12 months prior to screening
* Female participants postmenopausal >1 year or surgically sterile
* Two representative and similar target lesions for the condition, each of 15-25 centimeters squared (cm^2), up to 50 cm^2 in surface area
* Target lesion severity score of 4-8 on a scale of 0 to 12, where, in the opinion of the Investigator, 0 equals no evidence of disease and 12 equals severe induration, erythema, scaling, and pruritus
* Prescription medications, if applicable, for chronic conditions allowed but must be on a stable regimen prior to and during the study; this is also applicable for dietary supplements and over-the-counter (OTC) drugs
* Participants able and willing to give informed consent

EXCLUSION CRITERIA

* Use of any, concomitant, topical treatment for psoriasis, excluding emollients
* Use of any, concomitant, systemic treatment for psoriasis, including ultraviolet radiation (UVR) light
* Evidence of significant hepatic, gastrointestinal, renal, respiratory, endocrine, hematological, neurological, psychiatric, musculoskeletal, rheumatologic, or cardiovascular system abnormalities
* Evidence of any clinically significant deviation from normal with respect to medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), or clinical laboratory determinations. If any participant has an abnormal clinical laboratory test finding that meets specified criteria, that participant will be re-tested by repeated blood draw and clinical laboratory assessment. If the abnormal test finding is confirmed, the participant will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Total Symptom Severity (TSS) at week 8. | 8 weeks

SECONDARY OUTCOMES:
Total Symptom Severity (TSS) at all other time points; Physician's Global Assessment (PGA); safety; pharmacokinetics (PK) | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eisai US Medical Services, Study Director — Eisai Inc.
Locations (12):
- United States (12):
  - Hot Springs, Arkansas
  - San Diego, California
  - Boise, Idaho
  - Champaign, Illinois
  - Clinton Township, Michigan
  - Fridley, Minnesota
  - Omaha, Nebraska
  - Carlstadt, New Jersey
  - Portland, Oregon
  - Austin, Texas
  - College Station, Texas
  - Lynchburg, Virginia